CLINICAL TRIAL: NCT03584477
Title: Rehabilitation Program With Robotic Assistance for the Improvement of Motor Performance and Functional Use of the Upper Limb in Subacute Hemiparetic. Multicenter Randomized Controlled Trial
Brief Title: Robotic Rehabilitation of the Upper Limb After a Stroke
Acronym: ROBOASSIST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because inclusion rate was not met. No inclusion in the last 11 months.
Sponsor: Clinique Les Trois Soleils (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-A00632-39
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Stroke
Keywords: Stroke; Robot,; Rehabilitation; Hemiparesis; Upper limb; Function; Motor control
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional rehabilitation (Active Comparator): 5 sessions / week of 1 hour of occupational therapy
  Interventions: Other: Conventional rehabilitation
- Robotic rehabilitation with assistance (Active Comparator): 5 sessions / week of 1 hour of rehabilitation of the upper limb with 30 min of conventional rehabilitation and 30 min of robotic rehabilitation with assistance.
  Interventions: Device: Robot InMotion 2.0; Other: Conventional rehabilitation
- Non-assistance robotic rehabilitation (Active Comparator): 5 sessions / week of 1 hour of rehabilitation of the upper limb including 30 min of conventional rehabilitation and 30 min of robotic rehabilitation without assistance.
  Interventions: Device: Robot InMotion 2.0; Other: Conventional rehabilitation

INTERVENTIONS:
Device: Robot InMotion 2.0 — Repetitive work of large numbers of targeted alternative movements with or without assistance. The passage between with and without assistance taking place according to the evolution of performance judged by the investigator therapist. Note that the duration of the training using the assisted mode should be at least 3 weeks, i.e. half of the total duration of treatment.
  Arms: Non-assistance robotic rehabilitation; Robotic rehabilitation with assistance
Other: Conventional rehabilitation — Conventional rehabilitation implemented by an occupational therapist, involving stretching movements in submaximal passive amplitude, inhibition postures (Bobath), active efforts assisted of varied difficulty, exercises of direction of the arm towards a target with or without elbow support and grasping tasks, adapted to the capacities of the paretic upper limb.

SUMMARY:
Hemiparesis is the most common motor disorder after a stroke. Most patients do not recover functional use of their paretic upper limb.

The use of robotic assistance provides intensive motor training through a large number of repetitive movements, usually oriented and interactive tasks (pointing tasks, tracking paths tasks...). These feature have been demonstrated to be critical to stimulate brain plasticity after a brain damage. The InMotion Arm 2.0 manipulator works with an adaptive algorithm that provide patients with real-time Assistance-as-Needed™ desgned to enhance motor performance.

Hypothesis: In the sub-acute phase of stroke, the structured practice of a large number of repeated movements will increase motor function of the upper limb compared to conventional rehabilitation. Secondly, this practice will be more effective in a free active mode (without assistance) than an active assisted mode (Assistance-as-Needed™).

Expected secondary benefits: Subjective impression of improved use of the upper limb in activities of daily living and reduction of spastic cocontractions affecting the agonist and antagonist muscles during movements of the upper limb.

Objectives: This randomized controlled trial will evaluate the effects of structured repetition programs of arm movements, on the function of the hemiparetic upper limb and motor control, between 4 and 10 weeks after the stroke, using a robotic device with or without assistance in partial substitution of conventional rehabilitation care, compared to a program with conventional care alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Stroke hemiparesis on unilateral focal lesion dating from 4 to 10 weeks at baseline;
* Active flexion of the paretic shoulder ≥15 °;
* Average score on the modified scale of Frenchay <5;
* Patient having agreed to sign an informed consent.

Exclusion Criteria:

* Passive extension of the paretic elbow <120 °;
* Passive extension of the paretic wrist <10 °;
* Cognitive dysfunction or progressive intercurrent illness making effective communication or participation in the study impossible;
* Infection, inflammation or complex regional pain syndrome of the paretic upper extremity;
* Injection of botulinum toxin to the upper limb less than 3 months old;
* Patient under safeguard of justice;
* Patient include in an other clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Functional performance score change on Modified Frenchay Scale | Between the pre-rehabilitation state on the day of program start (Day1) and the state at the end of the program (Week6)
  The scale measures active upper limb function in hemiparesis based on 10 everyday living tasks, each rated on a 10-point visual analogic scale. Six tasks are bimanual and four are unimanual performed with the paretic hand. Final score is an average of the 10 subscores (10 is the higher score).

SECONDARY OUTCOMES:
Functional performance score change on Modified Frenchay Scale | between Day1 (day of program start) and Week22 (16 weeks after the end of the program)
  The scale measures active upper limb function in hemiparesis based on 10 everyday living tasks, each rated on a 10-point visual analogic scale. Six tasks are bimanual and four are unimanual performed with the paretic hand. Final score is an average of the 10 subscores (10 is the higher score).
Change of motor performance score on the Fugl-Meyer score | between Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
  Fugl-Meyer (FM) assessment for measures of the motor impairment of the upper-limb; the test includes items related to movements of the shoulder, elbow, forearm (proximal arm), and wrist and hand (distal arm). The total scores range between 0 and 66.

OTHER OUTCOMES:
Change in perceived function score on the Disability Assessment Scale (DAS) | between Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
  The scale evaluates upper limb functional disability in patients with spasticity following stroke. Patients are interviewed to determine the extent of functional impairment for the following 4 areas: hygiene,dressing, limb position, pain.The DAS Scale uses a 4-point rating scale according to the following criteria: 0(no disability),1 (mild disability), 2 (moderate disability) and 3(severe disability).
Change in perceived function score on the Global Subjective Self Assessment (GSSA) | between Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
  Three questions were asked to the patient, relating to pain, stiffness-induced discomfort and active function. Each rating was registered by the patient using a visual analogue scale ranging from 0 (worst pain imaginable, worst discomfort imaginable, arm totally useless, respectively) to 10 (no pain, no stiffness-induced discomfort, normal function, respectively).
Angle and grade of spasticity of the shoulder extensors, flexors and elbow pronators, clinically measured by the Tardieu modified scale | at Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
  The scale is a clinical measure of muscle spasticity for use with patients with neurological conditions. Spasticity is quantified by assessing the muscle's response to stretch applied at given velocities.
Paresis angle of shoulder flexion, extension and supination of the elbow; | at Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
  Paresis angle of shoulder flexion (maximal passive amplitude - maximal active amplitude)
Kinematic data of the movements based on the robot's records | at Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)
Maximum motor force measured by the robot of the abductor/adductor and flexors/extensors of the shoulder | at Day1(day of program start), Week6(end of the program) and Week22 (16 weeks after the end of the program)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Duret, MD, Principal Investigator — Clinique Les Trois Soleils; Jean-Michel Gracies, Pr, Principal Investigator — Hôpitaux Universitaires Henri Mondor
Locations (2):
- France (2):
  - Clinique Les Trois Soleils, Boissise-le-Roi
  - Hôpitaux Universitaires Henri Mondor, Créteil

IPD SHARING:
Plan to Share IPD: No